CLINICAL TRIAL: NCT00987870
Title: A Proof of Concept Study to Evaluate the Safety, Tolerability, and Pharmacodynamics of Multiple Topical Administrations of BFH772 in Patients With Psoriasis.
Brief Title: Safety and Efficacy of BFH772 in Psoriasis Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: CBFH772A2201; EUDRACT No. 2008-002795-96
Record Dates: First submitted 2009-09-30; First posted 2009-10-01 (Estimated); Last update posted 2011-03-28 (Estimated); Status verified 2011-03

CONDITIONS: Psoriasis; Arthritis
Keywords: Stable plaque Psoriasis; inflammatory skin; with or without arthritis
MeSH Terms: conditions — Psoriasis; Arthritis | interventions — calcipotriene; Betamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (5):
- BFH772 cream 1% (Experimental)
  Interventions: Drug: BFH772
- Placebo to BFH772 cream 1% (Placebo Comparator)
  Interventions: Drug: Placebo
- BFH772 ointment 1% (Experimental)
  Interventions: Drug: BFH772
- Placebo to BFH772 ointment (Placebo Comparator)
  Interventions: Drug: Placebo
- calcipotriol/betamethasone ointment (Active Comparator)
  Interventions: Drug: calcipotriol/betamethasone

INTERVENTIONS:
Drug: BFH772
  Arms: BFH772 cream 1%
Drug: Placebo
  Arms: Placebo to BFH772 cream 1%
Drug: BFH772
  Arms: BFH772 ointment 1%
Drug: Placebo
  Arms: Placebo to BFH772 ointment
Drug: calcipotriol/betamethasone
  Arms: calcipotriol/betamethasone ointment

SUMMARY:
This study will determine the efficacy of topical BFH772 in psoriasis patients and the safety after multiple dosing.

ELIGIBILITY:
Inclusion Criteria:

* Stable mild to moderate plaque psoriasis (BSA involvement < 10% or PASI < 10
* Category "mild to moderate" on PGA as according to the EMEA (CHMP 2004) (Guideline on clinical investigation of medicinal products indicated for the treatment of psoriasis), with or without arthritis
* Diagnosed or history of psoriasis for at least 6 months prior to screening

Exclusion Criteria:

* Nonplaque forms of psoriasis
* Drug-induced psoriasis
* Current use of beta blockers
* Congestive heart failure (NYHA >III), QT interval >450msec or poorly controlled diabetes mellitus

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-09; Primary Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Measure: Plaque PASI score | 4 weeks

SECONDARY OUTCOMES:
Measure: Local tolerability | Time Frame: baseline (predose Day 1) and 1h, 3h, 6h after the morning dose, then before each application (morning and evening) until the morning application on Day 5 and then at each visit before the morning application, and at study completion
Measure: BFH772 concentration in plasma | Day 1: Pre-dose; 4h post dose.
Measure: BFH772 concentration in skin | Week 4

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigator Site, Berlin, Germany